CLINICAL TRIAL: NCT01182051
Title: A Pilot Study of Family-based Cognitive-behavioral Therapy for Treating Chronic Pediatric Headache/Migraine and Comorbid Anxiety
Brief Title: A Study of Family-based Cognitive-behavioral Therapy for Chronic Pediatric Headache and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Migraine Research Foundation (Other)
Responsible Party: Principal Investigator, Golda S. Ginsburg, Ph.D., Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NA-00019444
Record Dates: First submitted 2010-05-21; First posted 2010-08-16 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2013-05

CONDITIONS: Pediatric; Headache; Anxiety
Keywords: headache; anxiety; pediatric headache and anxiety
MeSH Terms: conditions — Headache; Anxiety Disorders | interventions — Relaxation Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive behavioral therapy (Experimental): Key treatment ingredients in CBT include psychoeducation, trigger identification, progressive muscle relaxation training, cognitive restructuring, problem solving, in vivo exposure, and relapse prevention (see Appendix I for an outline of the treatment manual).
  Interventions: Behavioral: CBT or relaxation training
- Relaxation Training (Active Comparator): RT will consist of progressive muscle relaxation training, diaphragmatic breathing, and thermal biofeedback.
  Interventions: Behavioral: CBT or relaxation training

INTERVENTIONS:
Behavioral: CBT or relaxation training — 8 weeks of CBT or relaxation training.

SUMMARY:
The primary aim of this proposal is to refine the intervention under investigation (i.e., family-based CBT) and evaluate the feasibility and acceptability of the intervention and methods (e.g., recruitment, assessments).

The secondary aim of this proposal is to compare the relative efficacy of an 8 session family-based cognitive-behavioral therapy (CBT) to Relaxation Training (RT) for reducing anxiety and chronic headaches in youth (N = 30) ages 7-17 years. It is hypothesized that CBT will result in greater reductions in both anxiety and headache frequency and severity compared to RT.

DETAILED DESCRIPTION:
Chronic daily headache in children, as well as periodic migraine, is a prevalent, persistent, and debilitating pain condition affecting nearly 1 in 10 children. Emerging evidence suggests that affected youth also experience excessive and impairing symptoms of anxiety which may play a role in the etiology and/or maintenance of headache pain. Current behavioral treatments are effective in reducing headache frequency and intensity, however, many youth remain symptomatic and the exacerbating role of anxiety has largely been ignored. Moreover, current psychosocial treatments fail to incorporate parents in the therapeutic process. The current proposal is a pilot study designed to address the shortcomings of current behavioral treatments by evaluating the initial efficacy of a family-based cognitive-behavioral therapy (CBT) for youth who present with chronic tension headaches and migraines, and excessive anxiety. Rigorous scientific methods will be employed, including a randomized design, multiple informants and measures to assess key constructs, independent evaluators (IEs) to assess outcomes, and intensive training for therapists and IEs to assure a high quality of implementation. Using a pre-post experimental design, 30 youth with chronic tension headaches and/or migraines and anxiety will be randomly assigned to receive 8 weeks of family-based CBT or relaxation training (RT). IEs will complete assessments of child symptoms and functioning at pre and post-treatment and at one month follow-up. Youth in the family-based CBT condition are expected to evince greater reductions in both headache and anxiety frequency, severity, and duration. Results from this study will be used to make empirically informed modifications to the CBT treatment manual in order to facilitate replication and dissemination of the interventions to clinicians and researchers.

ELIGIBILITY:
Inclusion Criteria:

* To determine eligibility, youth will complete an evaluation consisting of clinical interviews, self-, and parent-report measures.
* To be included in the study, all children must:

  1. have a current diagnosis of chronic daily headache, tension-type headache, and/or migraine headache
  2. obtain a total score on the Screen for Child Anxiety Related Disorders (SCARED) in the clinical range (i.e., > 20)
  3. be between 7 and 17 years old
  4. have a parent/guardian who gives consent and agrees to participate
  5. be English speaking
  6. not currently participating in other psychosocial treatments specifically directed at reducing head pain or anxiety.
* For youth receiving prophylactic medication, it is preferable that they remain on a stable dose and agree to avoid medication changes while enrolled in the study. Thus, all participants will be permitted to continue with their prescribed medical/neurological treatment, however the use of medications (both prophylactic and over-the-counter analgesics) will be closely monitored.

Exclusion Criteria:

* Youth will be excluded from the study if they have a medical or psychiatric condition contraindicating study treatment or warranting an alternative intervention (e.g., suicidality, depression).

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2010-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Daily Headache and Anxiety Diary | Daily for three months
  Youth and parents will complete a daily headache and anxiety diary to track the frequency and severity of headaches and anxiety symptoms. In addition, the diary will assess medication use, missed school/activities, as well as antecedents and consequences.
Pediatric Anxiety Rating Scale (PARS) | 2 months
  The Pediatric Anxiety Rating Scale (PARS) will be completed by an independent evaluator to assess the severity of current (within the past week) anxiety symptoms in youth. The instrument consists of two sections. The first section contains a 50-item anxiety symptoms checklist. The second section assesses the severity and impairment of these symptoms. A total score is computed by summing the severity items. The measure has acceptable internal consistency, reliability, and convergent/divergent validity.

SECONDARY OUTCOMES:
Pediatric Migraine Disability Assessment (PedMIDAS) | 2 months
  The Pediatric Migraine Disability Assessment (PedMIDAS) is used to assess migraine disability across multiple domains of functioning including school, home, social, and recreational. The measure consists of 6 items measuring the number of days in which activities were missed as a result of headache/migraine. The measure yields a total score by summing items. Total scores correspond to one of four "disability grades:" 0-10 = little to no disability, 11-30 = mild disability, 31-50 = moderate disability, and >50 = severe disability.
Pediatric Migraine Disability Assessment (PedMIDAS) | 3 months
  The Pediatric Migraine Disability Assessment (PedMIDAS) is used to assess migraine disability across multiple domains of functioning including school, home, social, and recreational. The measure consists of 6 items measuring the number of days in which activities were missed as a result of headache/migraine. The measure yields a total score by summing items. Total scores correspond to one of four "disability grades:" 0-10 = little to no disability, 11-30 = mild disability, 31-50 = moderate disability, and >50 = severe disability.
Pediatric Anxiety Rating Scale (PARS) | 3 months
  The Pediatric Anxiety Rating Scale (PARS) will be completed by an independent evaluator to assess the severity of current (within the past week) anxiety symptoms in youth. The instrument consists of two sections. The first section contains a 50-item anxiety symptoms checklist. The second section assesses the severity and impairment of these symptoms. A total score is computed by summing the severity items. The measure has acceptable internal consistency, reliability, and convergent/divergent validity.

CONTACTS AND LOCATIONS:
Overall Officials: Golda S Ginsburg, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins, Baltimore, Maryland, United States